CLINICAL TRIAL: NCT02733549
Title: Is The Sudden Onset of Dizziness A Symptom of Acute Liver Dysfunction?An ED Study
Brief Title: Is The Sudden Onset of Dizziness A Symptom of Acute Liver Dysfunction?
Status: Completed | Type: Observational
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Umut Gulacti, principal investigator, Adiyaman University Research Hospital
Other Study IDs: ADYU-4
Record Dates: First submitted 2016-03-27; First posted 2016-04-11 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Dizziness
MeSH Terms: conditions — Dizziness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patient: Patients with sudden onset dizziness (SOD) analysed LFTs
  Interventions: Other: LFTs
- control: The control group with 98 healthy volunteer analysed LFTs
  Interventions: Other: LFTs

INTERVENTIONS:
Other: LFTs — A single 5-ml peripheral venous blood sample was collected from each participant.
  Serum ALT, AST, ALP, GGT, total bilirubin, conjugated bilirubin, and albumin level, Platelet count, INR and aPTT were analyzed.
  Other Names: liver function tests

SUMMARY:
Dizziness is one of the most common complaints among patients admitted to the emergency department (ED). In most cases, the etiology remains unclear. Dizziness has a broad differential diagnosis. The initial symptoms of ALD can include many general complaints. Aim of this study is to investigate whether SOD is a symptom of ALD, the necessity of liver function tests for patients with SOD in the ED, and a cost analysis of liver function tests.

DETAILED DESCRIPTION:
Dizziness is one of the most common complaints among patients admitted to the emergency department (ED). In most cases, the etiology remains unclear. Dizziness has a broad differential diagnosis. The initial symptoms of ALD can include many general complaints. The diagnosis of acute liver dysfunction (ALD) can usually be made by initial symptoms, physical examination, and biochemical tests, including liver function tests (LFTs) with high sensitivity and specificity. LFTs include albumin, bilirubin, coagulation factors (Activated Partial Thromboplastin Time (aPTT) and International Normalized Ratio (INR)), and liver enzymes, such as alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphates (ALP), and y-glutamyl transpeptidase (GGT), which are marker of hepatic damage. Aim of this study is to investigate whether SOD is a symptom of ALD, the necessity of LFTs for patients with SOD in the ED, and a cost analysis of LFTs.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients who were experiencing sudden onset dizziness of unknown etiology for the first time were included in the study

Exclusion Criteria:

1. Patients with a history of chronic diseases such as any liver disease,diabetes mellitus, hypertension,congestive heart failure, hepatitis B or C infection
2. Patients with any central dizziness attacks
3. Patients with hemodynamically unstable and emesis;
4. Patients receiving drugs that could affect liver function tests, such as, acetaminophen, antibiotics, oral contraceptives, antihypertensive drugs (e.g., angiotensinconverting enzyme inhibitors), or hormones (e.g.,estrogen)
5. Patients who was experienced dizziness with systemic diseases
6. Patients with any neurological disorders
7. Patient who do not want to participate in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult patients with sudden onset dizziness admitted to emergency department.
Sampling Method: Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
LFTs serum levels by biochemical method ALT, AST, ALP, GGT, total bilirubin, conjugated bilirubin, albumin, INR, aPTT, and Platelet count (PC) | 5 months
  The serum levels of LFTs will obtained by the laboratory analysis of blood samples of each participant.

SECONDARY OUTCOMES:
The cost calculation for the LFTs | 5 months
  The cost for the LFTs will be calculated with financial data in invoices which will obtained from the hospital invoicing service.

CONTACTS AND LOCATIONS:
Overall Officials: Umut Gulacti, Principal Investigator — Adiyaman University Medical Faculty
Locations (1):
- Adiyaman University Research Hospital, Adıyaman, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Giannini EG, Testa R, Savarino V. Liver enzyme alteration: a guide for clinicians. CMAJ. 2005 Feb 1;172(3):367-79. doi: 10.1503/cmaj.1040752. PMID 15684121
- [Background] Newman-Toker DE, Hsieh YH, Camargo CA Jr, Pelletier AJ, Butchy GT, Edlow JA. Spectrum of dizziness visits to US emergency departments: cross-sectional analysis from a nationally representative sample. Mayo Clin Proc. 2008 Jul;83(7):765-75. doi: 10.4065/83.7.765. PMID 18613993